CLINICAL TRIAL: NCT02267109
Title: A Phase 1b, Dose-escalating Safety and Immunogenicity Trial of the Novel Monovalent Ebola Zaire Candidate Vaccine, cAd3-EBO Z and the Heterologous Prime-boost Candidate Vaccine Regimen of cAD3-EBO Z Followed by MVA-BN® Filo in Malian Adults Aged 18-50 Years.
Brief Title: Phase 1 Trial of Ebola Vaccine in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Wellcome Trust (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Leidos Biomedical Research, Inc. (Industry)
Responsible Party: Principal Investigator, Milagritos Tapia, Assistant Professor, Pediatrics & Infectious Tropical Diseases, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HP-00061513
Record Dates: First submitted 2014-10-03; First posted 2014-10-17 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Ebola Virus Disease; Hemorrhagic Fever
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 2.5 x 10(10) vp (Experimental): Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z) 2.5 x 10(10):
  Interventions: Biological: Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z; Biological: Booster-MVA-BN® Filo or saline placebo
- 5 x 10(10) vp (Experimental): Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z) 5 x 10(10):
  Interventions: Biological: Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z; Biological: Booster-MVA-BN® Filo or saline placebo
- 1.0 x 10(10) vp (Experimental): Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z) 1.0 x 10(10):
  Interventions: Biological: Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z; Biological: Booster-MVA-BN® Filo or saline placebo
- 1.0 x 10(11) vp (Experimental): Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z) 1.0 x 10(11):
  Interventions: Biological: Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z; Biological: Booster-MVA-BN® Filo or saline placebo
- Booster-MVA-BN® Filo or saline placebo (Experimental): MVA-BN® Filo or saline placebo
  Interventions: Biological: Booster-MVA-BN® Filo or saline placebo

INTERVENTIONS:
Biological: Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z — IM injection of Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO Z):
  Other Names: cAd3-EBO Z:
  Arms: 1.0 x 10(10) vp; 1.0 x 10(11) vp; 2.5 x 10(10) vp; 5 x 10(10) vp
Biological: Booster-MVA-BN® Filo or saline placebo — IM injection of Booster-MVA-BN® Filo or saline placebo

SUMMARY:
Ebola virus causes an infection known as Ebola virus disease (EVD). This is generally a severe disease which can also lead to death. The 2014 outbreak of EVD in West Africa is the largest ever. Researchers want to develop a vaccine to prevent Ebola infection. It is impossible for someone to get an Ebola infection from this vaccine.

DETAILED DESCRIPTION:
This is a Phase 1b (1b implies that the trial is occurring in a geographic region where cases of the disease against which the vaccine is directed, i.e. Ebola disease, may occur before, during or after the clinical trial), open label, dose-escalation study to examine the safety, tolerability and immunogenicity of an investigational Ebola virus vaccine, cAD3-EB) Z, in Malian healthy adults. The vaccine is a recombinant chimpanzee adenovirus Type-3 vectored Ebola Zaire vaccine (cAd3-EBO Z) and consists of a recombinant replication-deficient adenovirus chimpanzee serotype 3 (cAd3) vector expressing wild-type (WT) Ebola glycoprotein (GP) from the Zaire strain.

A revision of the protocol on 14Dec2014 added a booster dose with MVA-BN® Filo or placebo in 56 subjects in groups 1 (except for first 5 vaccines), 2, 3A and 4. The multivalent vectored vaccine MVA-BN® Filo contains an insert for the Zaire Ebola virus glycoprotein, as well as the Sudan strain Ebola virus glycoprotein, the Musoke strain Marburg virus glycoprotein, and a nucleoprotein from the Tai-Forest Ebola virus.

Forty volunteers will be enrolled into two dosage groups. Another group of 40 volunteers (Groups 3A-C) with group 3A receiving 1.0x10(10)vp. All study participants will receive one dose of the study vaccine by intramuscular injection. Group 4 was added to include another 11 volunteers to receive 1.-X10(11)vp. A total of 91 volunteers have been included.

Group 1 will include 20 participants who will receive the lower dose of the vaccine at 2.5 x 10(10) vp

Group 2 will include 20 participants who will receive the higher does of vaccine at 5 x 10(10) vp.

Group 3A will include 10 participants to receive 1.0X10(10) vp

Group 3B will include 15 participants to receive 2.5X10(10) vp

Group 3C will include 15 participants to receive 5X10(10) vp (participants will be randomly allocated to Group 3B or 3C)

Group 4 will include 11 participants to receive1x10(11) vp. The goal of vaccinating this group is to see if there is any added benefit to the immunogenicity of this vaccine by using a higher dose. This dosage level of the monovalent vaccine has already been studied at VRC/NIH in September and at CVD in Baltimore this month in November. This dosage level was not studied in Oxford nor in Bamako. Having data on West African subjects given this dosage will be very helpful in designing the final formulation for the field trials in Q1 of 2015. The decision will be made based on three sets of data: clinical dose-response; immunologic dose-response (as a proxy for expected protection); and manufacturing yield and cost of goods considerations.

For safety reasons, the first Malian volunteer to receive a vaccine dose in Group 1 will be vaccinated alone and we will wait 24 hours before vaccinating subsequent volunteers in this dose group. Two further Group 1 volunteers may be vaccinated 24 hours after the first, and then at least another 24 hours gap will be left before vaccinating further subjects receiving that dose of vaccine. After 5 volunteers in Group 1 have been vaccinated and followed up for 7 days, an interim safety review (ISR1) will be performed by the DSMB. Enrollment of the rest of this group may proceed only if the DSMB assesses the data and indicates that it is safe to do so.

Group 2 volunteers will be vaccinated without the stepwise procedure. This decision was made by the DSMB after review of safety data for 5X10(10) from the UK trial and approval by the Institutional Review Boards.

Group 3A, who will receive a lower dosage level than Groups 1 or 2, can be vaccinated as soon as logistically possible after all subjects in Group 2 have been vaccinated. Groups 3B and Group 3C will be similarly vaccinated over a period of three days at the rate of 10 subjects per day.

Group 4 will vaccinate and additional 11 participants with 1X10(11) and will be vaccinated over 2 days (5 subjects one day followed by another 6 subjects the next day.

Heterologous boosting dose of MVA-BN® Filo or placebo in 56 subjects in groups 1 (except for first 5 vaccinees), 2, 3A and 4 will commence in January 2015 with random allocation to either vaccine or placebo.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults aged 18 to 50 years

* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with his/her health care provider
* For females only, willingness to practice continuous effective contraception (see section 6.4.3) during the study and a negative urine pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational Ebola or Marburg vaccine, a chimpanzee adenovirus vectored vaccine, MVA vectored vaccine or any other investigational vaccine likely to impact on interpretation of the trial data
* Receipt of any live, attenuated vaccine within 28 days prior to enrolment
* Receipt of any subunit or killed vaccine within 14 days prior to enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including urticaria, respiratory difficulty or abdominal pain
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Poorly controlled asthma or thyroid disease
* Seizure in the past 3 years or treatment for seizure disorder in the past 3 years
* Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
* Any known history of cardiac disease
* Any other serious chronic illness requiring hospital specialist supervision
* Current anti-tuberculosis prophylaxis or therapy
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Travel to an Ebola or Marburg endemic region during the study period or within the previous six months or history of recovery from Ebola or Marburg virus disease.
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-04-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited local and systemic reactogenicity signs and symptoms | Daily for 7 days following each vaccination.
Occurrence of unsolicited adverse events | 28 days following the vaccination
Change from baseline for safety laboratory measures | 6 months for each volunteer
Occurrence of serious adverse events and incident chronic medical conditions | 6 months for each volunteer

SECONDARY OUTCOMES:
Antibody responses as measured by ELISA and neutralization assays | Day 1, 7, 14, 28, 90 and 180 after vaccination
T cell immune responses as measured by intracellular cytokine staining assay | Day 1, 7 and 14 after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Myron M Levine, MD, DTPH, Study Director — University of Maryland, Baltimore
Locations (1):
- Center for Vaccine Development, Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tapia MD, Sow SO, Lyke KE, Haidara FC, Diallo F, Doumbia M, Traore A, Coulibaly F, Kodio M, Onwuchekwa U, Sztein MB, Wahid R, Campbell JD, Kieny MP, Moorthy V, Imoukhuede EB, Rampling T, Roman F, De Ryck I, Bellamy AR, Dally L, Mbaya OT, Ploquin A, Zhou Y, Stanley DA, Bailer R, Koup RA, Roederer M, Ledgerwood J, Hill AVS, Ballou WR, Sullivan N, Graham B, Levine MM. Use of ChAd3-EBO-Z Ebola virus vaccine in Malian and US adults, and boosting of Malian adults with MVA-BN-Filo: a phase 1, single-blind, randomised trial, a phase 1b, open-label and double-blind, dose-escalation trial, and a nested, randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2016 Jan;16(1):31-42. doi: 10.1016/S1473-3099(15)00362-X. Epub 2015 Nov 4. PMID 26546548